CLINICAL TRIAL: NCT06888505
Title: Mitigating Anthracycline-Induced Cardiac Toxicity With Dapagliflozin: A Randomized, Double-Blind, Placebo-Controlled Trial of 10 mg Daily for Four Months
Brief Title: Dapagliflozin to Prevent Anthracycline-Induced Cardiotoxicity
Acronym: DAPA-AIC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hawler Medical University (Other)
Collaborators: University of Zakho (Unknown)
Responsible Party: Principal Investigator, Hakar abdulkareem saeed, Principal Investigator; PhD Candidate, Hawler Medical University; Lecturer, University of Zakho, Hawler Medical University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: HSaeed; Hawler Medical University (Other: REC NO.: Meeting Code: 7, Paper Code: 4 Date: 27/05/2024); Duhok Directorate of Health (Other: Ethics Committee NO.: 31072024-6-17 Date: 31/07/2024)
Record Dates: First submitted 2025-03-03; First posted 2025-03-21 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Anthracyclines-Induced Cardiotoxicity; Cardiotoxicity
Keywords: cardiotoxicity; Anthracycline-induced cardiotoxicity; Dapagliflozin; SGLT2 inhibitors; cardio-oncology; Cardiac biomarkers in chemotherapy; Heart failure in cancer patients
MeSH Terms: conditions — Cardiotoxicity | interventions — dapagliflozin

STUDY DESIGN:
Intervention Model Description: This study is a randomized, double-blind, placebo-controlled trial investigating the efficacy of Dapagliflozin in preventing chemotherapy-induced cardiotoxicity in cancer patients receiving anthracycline-based chemotherapy.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: This is a double-blind, placebo-controlled trial in which participants, care providers, investigators, and outcomes assessors are blinded to treatment allocation. Randomization and treatment allocation will be conducted through a centralized system, and placebo tablets will be matched to ensure blinding.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dapagliflozin Arm (Active Comparator): Participants in this arm received dapagliflozin 10 mg orally once daily in addition to their standard anthracycline-based chemotherapy regimen.
  Dapagliflozin was continued daily for four months (throughout the chemotherapy treatment period).
  The study evaluated its potential cardioprotective effects against anthracycline-induced cardiac toxicity using echocardiography, cardiac biomarkers, and safety monitoring.
  Interventions: Drug: Dapagliflozin (Forxiga)
- Control Arm (Placebo Comparator): Participants in this arm received a placebo tablet identical in appearance, dosage form, frequency, and duration to dapagliflozin.
  The placebo was administered orally once daily for four months, alongside the participant's standard anthracycline-based chemotherapy regimen.
  The placebo contained no active ingredients and served as the control to evaluate the cardioprotective efficacy of dapagliflozin.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Dapagliflozin (Forxiga) — Participants in the dapagliflozin arm received dapagliflozin 10 mg tablets, administered orally once daily for 4 months, in addition to their standard anthracycline-based chemotherapy regimen. This treatment was given continuously throughout the chemotherapy period to evaluate its cardioprotective effects against anthracycline-induced cardiac toxicity.
  Other Names: Farxiga
  Arms: Dapagliflozin Arm
Other: Placebo — Participants in the control arm received a placebo tablet identical in appearance, dosage form, frequency, and duration to dapagliflozin, but containing no active ingredients. The placebo was administered orally once daily for 4 months alongside the participant's standard anthracycline-based chemotherapy regimen and served as the control to evaluate the cardioprotective efficacy of dapagliflozin.
  Other Names: Inactive tablet
  Arms: Control Arm

SUMMARY:
Brief Summary Anthracyclines (e.g., doxorubicin) are effective anticancer agents but can cause dose-dependent, often irreversible cardiotoxicity via oxidative stress, mitochondrial dysfunction, and cardiomyocyte apoptosis. Trastuzumab is also associated with left-ventricular dysfunction, typically reversible. The original protocol planned cohorts for both drug classes; however, no trastuzumab patients were enrolled due to feasibility, and the final study focused exclusively on anthracycline-treated patients.

Dapagliflozin, a sodium-glucose cotransporter-2 (SGLT2) inhibitor approved for diabetes and heart failure, has cardioprotective properties beyond glycemic control (reduced oxidative stress, inflammation, and fibrosis). We evaluated whether dapagliflozin mitigates anthracycline-induced cardiotoxicity.

This randomized, double-blind, placebo-controlled trial enrolled 90 patients receiving anthracycline-based chemotherapy. Participants were randomized 1:1 to:

1. dapagliflozin 10 mg orally once daily for 4 months plus standard chemotherapy; or
2. matching placebo once daily for 4 months plus standard chemotherapy. Primary outcome: change in left ventricular ejection fraction (LVEF) and diastolic function (e.g., E/A ratio, e'/E/e', diastolic dysfunction grade) from baseline to 16 weeks after chemotherapy initiation, measured by echocardiography.

Secondary outcomes: Troponin I, NT-proBNP, Galectin-3, CA 15-3, renal indices (creatinine, BUN, eGFR), and incidence of symptomatic cardiac dysfunction (e.g., heart failure, arrhythmias, myocardial infarction). Safety events related to chemotherapy or dapagliflozin were recorded and graded by CTCAE.

Assessments were performed at two time points only-baseline (pre-chemotherapy) and 16 weeks after initiation of chemotherapy; adverse events were collected continuously through the 16-week study period.

If effective, dapagliflozin could represent a practical cardioprotective strategy for patients receiving anthracyclines, potentially improving cardiovascular outcomes without compromising cancer therapy.

DETAILED DESCRIPTION:
Background and Rationale Chemotherapy-induced cardiotoxicity is a significant concern in cancer treatment, particularly with anthracyclines (e.g., doxorubicin). Anthracycline-induced cardiotoxicity is often irreversible, resulting from oxidative stress, mitochondrial dysfunction, and direct cardiomyocyte apoptosis.

Trastuzumab (Herceptin) is another major cardiotoxic drug, though its effects are often reversible. The initial protocol was designed to include both anthracycline- and trastuzumab-treated patients. However, due to feasibility constraints, the trastuzumab cohort was not enrolled, and the final study focused solely on patients receiving anthracycline-based chemotherapy.

Dapagliflozin, a sodium-glucose co-transporter-2 (SGLT2) inhibitor, is primarily used for type 2 diabetes mellitus and heart failure with reduced ejection fraction (HFrEF). Emerging evidence suggests cardioprotective properties independent of glucose control, including:

Reduction of oxidative stress and myocardial fibrosis Improvement of mitochondrial efficiency and myocardial metabolism Reduction in systemic and myocardial inflammation Modulation of sodium and calcium handling in cardiomyocytes Given these mechanisms, dapagliflozin may provide a protective effect against anthracycline-induced cardiotoxicity, preserving cardiac function without compromising cancer treatment efficacy.

Study Design and Methodology This is a randomized, double-blind, placebo-controlled clinical trial designed to evaluate the cardioprotective effects of dapagliflozin in cancer patients undergoing anthracycline-based chemotherapy.

Study Sites Primary Location: Azadi Oncology Center affiliated with Hawler Medical University and the Duhok General Health Directorate.

Multicenter expansion was considered, but all participants were recruited at the primary site.

Study Population Enrollment (Actual): 90 participants receiving anthracycline-based chemotherapy.

Randomization ratio: 1:1 (45 patients per group). Intervention and Control Groups Control Group (n=45): Standard chemotherapy + placebo. Dapagliflozin Group (n=45): Standard chemotherapy + dapagliflozin (10 mg/day, oral) for four months.

Follow-up Period Duration: 4 months from initiation of chemotherapy. Assessment intervals: Baseline (pre-chemotherapy) and 4 months (post-chemotherapy completion).

Primary outcome: Change in left ventricular ejection fraction (LVEF) and diastolic function-assessed by transmitral E/A ratio, average septal/lateral e', E/e', and graded per ASE/EACVI criteria-from baseline to 16 weeks after chemotherapy initiation, measured by echocardiography.

Secondary Endpoints Cardiac Biomarkers: Troponin I, NT-proBNP, Galectin-3. Cancer Progression Marker: CA 15-3. Renal Function: Creatinine, BUN, eGFR. Adverse Events: Incidence of chemotherapy- and dapagliflozin-related adverse effects, graded per CTCAE.

Safety and Monitoring Plan Echocardiography: Baseline and 4 months. Biomarkers: Baseline and 4 months. ECG: Performed if clinically indicated to detect arrhythmias or QT prolongation.

Adverse Events: Monitored continuously throughout the 4-month treatment and follow-up, including risks of hypoglycemia, hypotension, dehydration, renal events, urinary tract infections, and ketoacidosis.

Statistical Analysis Plan Sample Size: Originally planned for 100 patients, but 90 were enrolled (45 per group).

Comparative Analysis: Paired t-tests, Wilcoxon signed-rank tests (for non-parametric data), ANOVA for repeated measures where appropriate.

Multivariate Regression: Adjusting for age, baseline cardiac function, and cumulative anthracycline dose.

Missing Data: Addressed using multiple imputation to maintain robustness. Ethical Considerations Approved by Hawler Medical University Ethics Committee and the Duhok General Health Directorate.

Written informed consent obtained from all participants. Potential Impact If dapagliflozin proves effective, this study could support the use of SGLT2 inhibitors as a cardioprotective strategy in anthracycline-treated cancer patients, improving cardiovascular outcomes, long-term survival, and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed breast cancer (or other cancers as relevant to the study).
* Age 18-70 years.
* Planned treatment with anthracycline-based chemotherapy
* Normal kidney function, defined as serum creatinine 0.6-1.2 mg/dL.
* Normal liver function, defined as ALT and AST 10-40 U/L.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-2.
* Willingness to participate and provide written informed consent.

Exclusion Criteria:

* History of symptomatic heart failure (NYHA class III-IV) or prior anthracycline-related cardiac dysfunction.
* Previous use of Dapagliflozin.
* Pregnancy or breastfeeding.
* Severe renal impairment (eGFR < 30 mL/min/1.73m²).
* Uncontrolled diabetes mellitus (HbA1c > 9%).
* Active or recurrent urinary tract infections (UTIs) within the last 6 months.
* Known hypersensitivity to Dapagliflozin or related compounds.
* Concurrent participation in another clinical trial investigating cardioprotective agents.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2024-09-01 (Actual); Primary Completion 2025-09-01 (Actual); Study Completion 2025-09-06 (Actual)

PRIMARY OUTCOMES:
Left Ventricular Function (Systolic and Diastolic) | Evaluated at baseline and 4 months after initiation of chemotherapy.
  Echocardiographic assessment of left ventricular systolic function (LVEF) and diastolic function (E/A ratio, diastolic dysfunction grade) to detect anthracycline-induced cardiotoxicity.Measurement Tool: Echocardiography (using a 2D echocardiogram).

SECONDARY OUTCOMES:
Cardiac Troponin I Levels | Evaluated at baseline and 4 months after initiation of chemotherapy.
  Measurement of serum Troponin I levels to assess myocardial injury and cardiac stress in patients undergoing chemotherapy.
  Measurement Tool: Chemiluminescent Immunoassay (CLIA).
NT-proBNP Levels | Evaluated at baseline and 4 months after initiation of chemotherapy.
  Measurement of serum NT-proBNP levels as an indicator of cardiac stress and dysfunction.
  Measurement Tool: Chemiluminescent Immunoassay (CLIA).
Galectin-3 Levels | Evaluated at baseline and 4 months after initiation of chemotherapy.
  Measurement of serum Galectin-3 levels to evaluate its role in oxidative stress, apoptosis, and tissue remodeling.
  Measurement Tool: Enzyme-Linked Immunosorbent Assay (ELISA).
CA 15-3 Levels | Evaluated at baseline and 4 months after initiation of chemotherapy.
  Measurement of serum CA 15-3 levels to monitor breast cancer cell proliferation.
  Measurement Tool: Chemiluminescent immunoassay
Kidney Function Tests | Evaluated at baseline and 4 months after initiation of chemotherapy.
  Monitoring of serum creatinine and blood urea nitrogen (BUN) to assess renal function and potential nephrotoxicity related to chemotherapy or Dapagliflozin.
  Measurement Tool: Automated Biochemical Analyzer for serum creatinine and BUN.
Complete Blood Count (CBC) | Evaluated at baseline and 4 months after initiation of chemotherapy.
  Monitoring of hematological parameters (e.g., hemoglobin, white blood cells, platelets) to assess overall health, immune function, and tolerability of treatment.
  Measurement Tool: Automated Hematology Analyzer (Beckman Coulter analyzers).
Liver Function Tests (LFTs) | Evaluated at baseline and 4 months after initiation of chemotherapy.
  Monitoring of liver enzymes (e.g., ALT, AST, alkaline phosphatase, bilirubin) to assess liver function and potential hepatotoxicity due to chemotherapy or Dapagliflozin.
  Measurement Tool: Chemiluminescent Immunoassay

CONTACTS AND LOCATIONS:
Overall Officials: Hakar A Saeed, M.Sc, Principal Investigator — University of Zakho; Nidhal A Mohammed Ali, PhD, Principal Investigator — Hawler Medical University; Ramadhan T Othman, PhD, Principal Investigator — University of Duhok
Locations (1):
- Azadi Oncology Centre, Duhok, Iraq

IPD SHARING:
Plan to Share IPD: No
At this time, individual participant data (IPD) will not be shared publicly. The data will be kept confidential to ensure participant privacy and comply with ethical and regulatory requirements, including those related to informed consent and data protection. Access to the data may be considered for future collaborations under strict ethical guidelines and approval from the relevant oversight bodies.